CLINICAL TRIAL: NCT00284752
Title: Phase II Trial of Abraxane in Front Line Therapy of Hormone Refractory Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TK001
Record Dates: First submitted 2006-01-30; First posted 2006-02-01 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Prostate Cancer
Keywords: Prostate; Cancer; Metastatic
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Neoplasm Metastasis | interventions — Albumin-Bound Paclitaxel

ARMS (1):
- ABI-007 (Experimental)
  Interventions: Drug: Abraxane

INTERVENTIONS:
Drug: Abraxane — This is a Phase II single-arm study for first-line chemotherapy of patients with hormone refractory metastatic prostate cancer. Eligible patients will be chemotherapy naive and will receive weekly Abraxane 100mg/m2 IV over 30 minutes. These will be 4-week cycles with patients receiving Abraxane 100 mg/m2 weekly for 3 weeks and one week off for rest. Patients will continue on therapy until disease or PSA

SUMMARY:
Evaluate the efficacy of Abraxane in first line chemotherapy of patients with hormone refractory metastatic prostate cancer, based on prostate specific antigen (PSA) response

DETAILED DESCRIPTION:
Taxanes are the most widely tested and effective chemotherapy drugs for hormone refractory prostate cancer. Weekly paclitaxel was reported to produce 25-39% PSA responses in first line and up to 33% in second line chemotherapy of patients with prostate cancer in early clinical trials (1, 2). Paclitaxel activity in prostate cancer is schedule dependent, and weekly paclitaxel was reported to produce highest response rates (1, 2). Docetaxel was recently approved by the Food and Drug Administration for treatment of hormone refractory metastatic prostate cancer, since it is the only chemotherapy drug with documented improvement in survival in this group of patients. Docetaxel was associated with 45.8% overall grade 3/4 toxicities and it has to be given with steroid pre-medication. This regimen might be difficult to use in advanced prostate cancer patients that are often elderly and with multiple co-morbid conditions.

ABI-007 [Abraxane™ (paclitaxel protein-bound particles for injectable suspension) (albumin-bound)] is the first in its class of biologically interactive albumin-bound forms of chemotherapy (3). This composition provides a novel approach of increasing intra-tumoral concentration of the drug by a receptor-mediated transport process allowing transcytosis across the endothelial cell wall, thereby breaching the blood/tumor interface. This albumin-specific receptor mediated process involves the binding of a specific receptor (gp60) on the endothelial cell wall, resulting in activation of a protein caveolin-1, which initiates an opening in the endothelial wall with formation of a little caves or caveolae, with transport of the albumin-bound chemotherapeutic complex via these caveolae to the underlying tumor interstitium (4). A protein specifically secreted by the tumor (SPARC) binds and entraps the albumin, allowing release of the hydrophobic drug to the tumor cell membrane. ABI-007 is the first biologically interactive albumin-bound chemotherapy agent leveraging this gp-60/caveolin-1/caveolae/Sparc pathway to increase intra-tumoral concentration of the drug and reduce the amount of the toxic chemotherapy in normal tissue.

Preclinical studies comparing Abraxane to paclitaxel demonstrated lower toxicities, with a maximum tolerated dose (MTD) approximately 50% higher for Abraxane (7) compared to paclitaxel (11). At equal doses there was less myelosuppression and improved efficacy than paclitaxel in a xenograft tumor model of human mammary adenocarcinoma. Clinical studies confirmed improved toxicity profile and higher response rates, in metastatic breast cancer, of Abraxane compared to cremophor EL paclitaxel (Taxol) (5, 8). The weekly regimen was shown to be active even in patients with cancers refractory to paclitaxel, docetaxel or when Abraxane was given after both agents (8).

ELIGIBILITY:
Inclusion Criteria:

1. Histopathologically or cytologically proven adenocarcinoma of the prostate metastatic to the bones or lymph nodes as documented by bone scan or CT scan with evidence of progression despite standard hormonal management (orchiectomy, GNRH agonist, or GNRH antagonist-hormone refractory). No major organ allowed
2. No prior chemotherapy
3. For patients who have been on anti-androgen therapy, patients must have progressive disease after anti-androgen withdrawal (6 weeks biclutamide or nilutamide, 4 weeks for flutamide).
4. PSA progression is defined as rising PSA.

Exclusion Criteria:

1. Active malignancy other than non-melanoma skin cancer within 5 years of enrollment.
2. Significant active medical illness which in the opinion of the investigator will preclude treatment.
3. Brain metastasis, any non-bone metastasis except lymph node metastasis

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2005-08; Primary Completion 2007-10 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of Abraxane in first line chemotherapy of patients with | August 2008
hormone refractory metastatic prostate cancer, based on prostate specific antigen (PSA) response | August 2008

SECONDARY OUTCOMES:
Evaluate the effect of Abraxane on,Time to PSA progression, Measurable tumor response rate (if measureable disease at baseline), Overall survival | August 2008
Evaluate the toxicity of Abraxane in this group of patients. | August 2008

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Kolevska, MD, Principal Investigator — Kaiser Permanente
Locations (1):
- Kaiser Permanente, Vallejo, California, United States